

# **ISGlobal - Barcelona Institute for Global Health**

"Expanding Xpert Ultra for TB diagnosis among HIV-positive patients admitted to hospitals in Tanzania and Mozambique (EXULTANT)"

# STATISTICAL ANALYSIS PLAN

Version 2.0 dated 06-December-22

Author/s: Sergi Sanz

Tel: Carrer Rosselló 132, 7a planta

E-08036 Barcelona, Spain

Tel. 034 932 275 400 ext. 2790

sergi.sanz@isglobal.org



**Protocol Number: TB043-3/1** 

# **Approval Page**

The signatures below confirm that the signatories have reviewed and approved this document which shall govern the stipulated statistical analysis tasks of the specified research study.

| Sergi Sanz | | Statistician (ISGlobal) |
|---|---|---|
| Name | SERGIO SANZ Firmado digitalmente por SERGIO SANZ BRAVO - DNI - DNI 44178555V Fecha: 2023.01.09 15:55:05 +01'00' | Designation |
| Signat | ure | Date |
| Stefano | o Ongarello | Reviewer (Director, Data Science) |
| Name | | Designation |
| Staf | igned by:<br>ans Ongarells | 1/17/2023 |
| Signat | 4FB108242C<br><b>ure</b> | Date |
| Berra E | Erkosar | Reviewer (Senior Statistician) |
| Name | | Designation |
| Docus | igned by: | 1/19/2023 |
| Signat | 63E503846D<br>Ure | Date |
| Vinzeig | jh Leukes | Trial Manager |
| Name | | Designation |
| Viwy | igned by:<br>Ligh Leukes | 1/17/2023 |
| Signat | 2EB4CF44F2<br><b>Ure</b> | Date |



# **Table of Contents** 2 2.1 Study Objectives and Endpoints ...... 6 Main Study Objectives ...... 6 3.1 3.2 Secondary and Exploratory Study Objectives ....... 6 3.3 Study design ...... 6 Study Methods ...... 8 4.1 General Study Design and Plan ...... 8 4.2 4.3 Randomisation and Blinding ...... 10 4.4 5 General Considerations 20 6.1 6.2 7 Summary of Study Data ......21 7.1 Subject Disposition......21 7.2 8.1 8.2



# **Statistical Analysis Plan**

| 9. | Subgroup analysis25 |
|-----|-----------------------------------------|
| 10. | Other Analyses |
| 11 | Reporting Conventions |
| 12 | Technical Details |
| 13 | Listing of Tables, Listings and Figures |



#### 1 Abbreviations and Definitions

| AE | Adverse Event |
|---|---|
| AlereLAM | Alere Determine TB LAM Ag |
| CRF | Case Report Form |
| DMP | Data Management Plan |
| FujiLAM | Fujifilm SILVAMP TB LAM |
| HIV | Human immunodeficiency virus |
| IMP | Investigational Medical Product |
| ITT | Intention to treat |
| KPS* | Karnofsky Performance Status Scale definitions rating (%) criteria |
| LF-LAM | Lateral flow urine lipoarabinomannan assay |
| PP | Per Protocol |
| SAP | Statistical Analysis Plan |
| TB | Tuberculosis |
| Ultra | Xpert MTB/RIF Ultra |

#### 2 Introduction

#### 2.1 Preface

Tuberculosis (TB) is a leading cause of death worldwide and ranks above HIV/AIDS as the leading cause of mortality from a single infectious agent. The World Health Organization (WHO) estimated that there were around 10 million new cases and 1.5 million deaths in 2021. Eight and 14% of the total number of TB cases and deaths respectively occurred in people living with HIV (PLHIV), with 70% of these occurring in the African region. PLHIV are at increased risk of acquiring Mycobacterium tuberculosis (Mtb) infection and have a >20-fold increased risk of TB disease progression compared to HIV-uninfected peers. In addition, mortality during TB treatment remains as high as 11% globally, although fatal outcomes of PLHIV under TB treatment are even higher in Sub-Saharan African countries

Among people living with HIV, microbiological confirmation of TB is suboptimal due to sputum collection challenges and paucibacillary sputum resulting in poor diagnostic yield. Options that have been recommended by WHO to ensure earlier diagnosis and reduce mortality include strategic placement of rapid molecular TB diagnostics such as Xpert or Ultra within HIV care settings (which could enable availability of results within 24 hours), and uptake of the urine lipoarabinomannan assay (LF-LAM) strip-test, the Alere Determine™ TB LAM Ag (AlereLAM), for seriously ill or immunosuppressed PLHIV. However, despite AlereLAM being a cheap and fast test, only 9 of the 30 high TB and HIV burden countries had in 2020 a national policy and algorithm indicating the routine use of urine LF-LAM (with various levels of implementation). In addition, PLHIV often are sputum paucibacillary and a considerable proportion of them cannot provide a good quality sputum specimen for molecular testing.



The limitations of existing sputum-based tests for M. tuberculosis (Mtb) diagnosis among (PLHIV) admitted to hospital create imperatives to explore the usefulness of easy to collect, non-respiratory specimens which could improve TB diagnosis, while supporting and accelerating treatment guidance. Previous studies have shown that Xpert testing of urine and stool can confirm Mtb in participants who would otherwise test negative with traditional sputum-based methods. Evidence shows that these diagnostics may detect additional cases that are not detected by AlereLAM. Thus, an algorithm using the different tests (sputum Ultra, urine Ultra and stool Ultra) offered as a screening intervention to admitted HIV positive participants should increase the Mtb bacteriological yield (compared to current WHO recommended screening and testing strategies\*\*) and contribute to earlier initiation of TB treatment. Given that some detected cases may not present with classical TB symptoms at the time of hospitalization, we believe that this strategy will increase the overall number of participants with diagnosed TB and started on treatment and ultimately reducing mortality.

## 3 Study Objectives and Endpoints

## 3.1 Main Study Objectives

The primary objective of the study is to investigate the effect of an expanded TB screening strategy performed in HIV-positive participants admitted to hospital on the proportion of bacteriologically confirmed TB cases starting treatment within 72 hours of enrolment

**INTERVENTION ARM** (expanded TB screening strategy): Xpert Ultra on sputum, stool/rectal swab and AlereLAM on urine, performed regardless of presence of TB symptoms

**CONTROL ARM**: Ultra testing (on sputum/any tissue) if TB-compatible symptoms and AlereLAM (on urine) only in those fulfilling WHO testing recommendations.

# 3.2 Secondary and Exploratory Study Objectives

The study has the following secondary objectives.

# Secondary objectives

- 1. To assess the impact of this screening strategy on 2-month all-cause mortality.
- 2. To assess the feasibility of multiple specimen collection for TB diagnosis within 72 hours of enrolment.

\*to the main protocol includes additional exploratory objectives, which will be specified in a separate SAP

### 3.3 Study design



This is a multicentre, parallel, individually randomized, controlled diagnostic trial in consecutively enrolled HIV positive adults admitted to hospital in selected sites in Mozambique and Tanzania.

This trial has two study arms, the intervention and control arm. The intervention arm for this study consists of HIV participants with TB testing performed regardless of presence of TB symptoms. Testing will be done on expectorated sputum, stool/rectal swab and concentrated urine with Ultra and urine with AlereLAM.

The <u>control arm</u> for this trial will consist of participants managed according to the current WHO recommended TB testing practices for HIV positive in participants (as of Q1 2022). TB testing will be done as follows:

**Sputum Ultra** performed whenever the patient has cough, fever, weight loss overnight sweats and/or

**Ultra performed on any tissue** (including lymph nodes) from participants with clinical suspicion of extrapulmonary TB.

#### and/or:

*Urine Alere TB-LAM* performed if participants have signs and symptoms of TB (pulmonary and/or extrapulmonary), or with advanced HIV disease, or who are seriously ill, or else irrespective of signs and symptoms of TB, but combined with a CD4 cell count of less than 200 cells/mm<sup>3</sup>.

## 3.4 Endpoints

All study endpoints will be compared between control and intervention arm. Also, the final results will be presented disaggregated by sex.

- 3.4.1 The **primary endpoint** is the proportion of participants diagnosed with microbiologically confirmed TB and started on TB treatment within 72 hours of enrolment\* in whom TB is microbiologically confirmed\*/\*\*
- \* The numerator of the primary endpoint includes participants per study arm who are diagnosed with microbiologically confirmed TB and initiated TB treatment within 72 hrs of enrolment. The denominator is the number of enrolled participants in each study arm.
- \*\* Participants are defined to have microbiologically confirmed TB if at least one confirmatory TB test (Ultra, AlereLAM) gives a positive result.

### Secondary endpoints are:

Related to main objective

- 3.4.2.1 Time-to-TB-treatment-initiation among microbiologically confirmed cases and among all TB cases since enrolment. We will estimate Kaplan Meier curves and hazard ratios at day 7, 14, 28 and 56. Additionally we will compare the time to related estimates (median and IQR) of intervention and control group.
- 3.4.2.2 Proportion of cases re-admitted to hospital. The numerator will be the number of admissions for any reason (not included in the exclusion criteria) after initial discharge and within 8 weeks from enrolment. The denominator will be the number of participants enrolled.



- 3.4.2.3 Proportion of participants who are diagnosed with TB (irrespective of bacteriological confirmation) and have started on TB treatment within 72 hours of enrolment.
- 3.4.2.4 Proportion of participants who are diagnosed with microbiologically confirmed TB and are started on treatment at 7, 14 days and 8 weeks of enrolment.
- 3.4.2.5 Time to laboratory confirmed TB diagnosis and any TB diagnosis since enrolment.
- 3.4.2.6 Proportion of microbiologically confirmed TB participants started on treatment without Rif resistance information (only AlereLAM positive)).

Related to secondary objectives.

- 3.4.2.7 Eight-week all-cause mortality. The numerator will be the number of deaths during eight weeks after enrolment, the denominator the number of participants enrolled.
- 3.4.2.8 In hospital and 4-week all-cause mortality among all participants enrolled (assessed as the eight-week all-cause mortality).
- 3.4.2.9 Proportion of study participants who are able to provide the different specimens (sputum and urine samples) within 24, 48 and 72 hours of enrolment in the control and treatment arms.

# 4 Study Methods

# 4.1 General Study Design and Plan

The study design is a multicentre, parallel, individually randomized, controlled diagnostic trial in consecutive HIV positive adults admitted to hospital in selected sites of Mozambique and Tanzania.

Schedule of Visits.



# **Statistical Analysis Plan**

| | Day 0<br>(recruitment<br>) | Day 0<br>(recruitment) | Day 0-3 | Daily | At discharge<br>If discharged<br>before day 28/56 | Week 4<br><u>+/- 3</u> | Week 8<br>days |
|---|---|---|---|---|---|---|---|
| Control arm | | Intervention arm | (<72h) | | | | |
| Baseline Evaluation | | | | | | | |
| Informed consent | X | Χ | | | | | |
| Eligibility criteria verified | X | Χ | | | | | |
| CD4 count / Viral Load <sup>&amp;</sup> | X | Χ | | | | | |
| Locator information | X | Χ | | | | | |
| Brief medical history | X | Χ | | | | | |
| Proof of HIV status stored | X | Χ | | | | | |
| WHO Symptom screening | X | Χ | | | Χ | | |
| TB Investigations Samples collected and tests Results issued | Urine<br>AlereLAM#<br>Sputum<br>Ultra*<br>Blood CD4 | Sputum Ultra Stool/rectal swab Ultra Urine Ultra Urine AlereLAM 2x Oral Swabs Urine FujiLAM Blood CD4 Blood for CRP | X | | | | |
| Further contacts | | | | | | | |
| Verification TB diagnosis / ad hoc TB investigations | | | | Х | Χ | X | Χ |
| Verification TB treatment initiation | | | | Х | Χ | Χ | Х |
| Verification vital status | | | | X | X | X | X |
| HIV care / ART | | | | X | X | X | X |



## 4.2 Inclusion-Exclusion Criteria and General Study Population

This study has the following inclusion and exclusion criteria.

#### Inclusion criteria:

- 1. Adults 18 years or older.
- 2. Confirmed HIV infection (including both antiretroviral (ART)-naïve and experienced).
- 3. Admitted to the hospital (adult medical wards) at the time of enrolment.

#### **Exclusion criteria:**

- 1. Unable to provide informed consent (if no authorized relatives are in the position to provide the consent).
- 2. Living outside the catchment area of the participating hospital(s).
- 3. With plans to migrate outside the catchment area within 2 months after recruitment.
- 4. Currently receiving anti-TB therapy or having received anti-TB therapy in the last 6 months prior to enrolment.
- 5. Receiving preventive TB treatment in the preceding 6 months
- 6. Participants admitted for traumatic reasons, acute abdomen, delivery or pregnancy (maternal conditions), or for planned/scheduled surgery.
- 7. Referred from other hospital
- 8. Positive result to a SARS-CoV-2 test (RT-PCR, antigen test, or other similar test that might define COVID-19 case in the study site)\*

# Study population

The study population will be adult (≥18 years) PLHIV participants admitted to hospital and living in the catchment areas within the 4 district hospitals in Tanzania and Mozambique, regardless of presence of TB compatible symptoms.

### 4.3 Randomisation and Blinding

This is an individually randomized clinical trial. Eligible participants will be randomized to either the intervention or control arm, with 50% of participants in each of the arms. Randomization will be conducted using a web-based application <a href="https://odk-central.finddx.org/-/x/6RPyVJQoEjzOPUd3qHIRQYX6MtFnnwq">https://odk-central.finddx.org/-/x/6RPyVJQoEjzOPUd3qHIRQYX6MtFnnwq</a> that can be used on any smartphone device with internet connection. The day of randomization for each participant will be the enrolment day (study Day 0). At the time a participant is randomized, the study staff enters in the application several key data (patient study number and date of birth) and in reply, the allocated randomized arm is provided a few seconds later in the same application interface. Thus, internet connection is needed for randomizing participants. Pre-registered users of the study team will be allowed to use the randomization application.



Developing a reliable training plan by which study teams (at the clinic and at the lab) are fully aware of the diagnostic allocation is critical so that arm-specific testing can be implemented without mistakes in a timely manner. This includes careful strategic measures (posters, signs, weekly meetings, etc) as part of the site internal planning, which also need to consider staff shifts, holidays (both in the hospital and at the laboratory). A screening and randomization log need to be daily updated. Day 0 CRF needs to be data entered in a timely manner to allow the central monitoring of number of recruited subjects per arm, site and week and overall mapping of participants included in the study.

This is an unblinded trial. Neither participants, nor study staff will be blinded to tests practiced or test results.

# 4.4 Study Variables

The Baseline participants variables we will collected from TB-CAPT-HIV EXULTANT-BaselineCharacteristics-v3, and the following versions of this document. From this CRF the important variables for the analysis are:

| Variable | | Used in |
|---|---|---|
| Label | name | J Good III |
| Date of enrolment | ENROL_D | To calculate endpoints related to time. |
| Time of enrolment | ENROL_T | To calculate endpoints related to time. |
| Country | COUNTRY | To adjust some regression models. For previous analysis about at random lost to follow up. |
| Sex | SEX | To describe the participant's profile. For previous analysis about at random lost to follow up. |
| Ethnic group | ETHNIC_SPEC | To describe the participant's profile. For previous analysis about at random lost to follow up. |



| | EDUCATION | To describe the participant's |
|---|---|---|
| | EDUCATION ODEO | profile. |
| Level of education | EDUCATION_SPEC | For previous analysis about at |
| | | random lost to follow up. |
| | EMPLOYMENT | To describe the participant's |
| | EMDLOVMENT SDEC | profile. |
| Employment Status | EMPLOYMENT_SPEC | For previous analysis about at |
| | | random lost to follow up. |
| Type of Employment: | EMPL_HLTH_YN | |
| 2.6 Is the patient employed as a | EMPL PRSN YN | |
| health care worker? | | To describe the participant's |
| 2.7 Is the patient employed as a | EMPL_MINE_YN | profile. |
| prison warder/work at a | | For previous analysis about at |
| correctional facility? | | random lost to follow up. |
| 2.8 Is the patient employed as a | | |
| miner? | | |
| Early HIV positive result | HIV_POS_DATE | To describe the participant's |
| 3.1.1 Date of earliest HIV | | profile. |
| positive result: | | For previous analysis about at random lost to follow up. |
| | | random lost to follow up. |
| | ART_YN | To describe the participant's |
| Current taking antiretroviral | | profile. |
| | | For previous analysis about at |
| | | random lost to follow up. |
| | TB_TX_YN | To describe the participant's |
| Previous TB episodes | | profile. |
| | | For previous analysis about at |
| | | random lost to follow up. |
| | BCG_YN | To describe the participant's |
| Received BCG vaccination | | profile. |
| | | For previous analysis about at |
| | | random lost to follow up. |



| Participant live alone? | CTX YN | To describe the participant's profile. For previous analysis about at random lost to follow up. To describe the participant's |
|---|---|---|
| Patient taking cotrimoxazole? | | profile. For previous analysis about at random lost to follow up. |
| High blood pressure | HIGH_RR_YN | To describe the participant's profile. |
| Diabetes | DIABETES_YN | To describe the participant's profile. |
| Cardiac disease | CARDIAC_YN | To describe the participant's profile. |
| Epilepsy | EPILEPSY_YN | To describe the participant's profile. |
| Karnofsky Performance Status<br>Scale | KARNOFSKY | To describe the participant's profile. For previous analysis about at random lost to follow up. |
| Patient's WHO clinical Stage | WHO_STAGES | To describe the participant's profile. For previous analysis about at random lost to follow up. |
| TB treatment start | TB_TX_START_YN | To describe the participant's profile. For previous analysis about at random lost to follow up. |
| Random group | RANDOM_ASSIGN | For previous analysis about at random lost to follow up. |
| Date of randomization | RANDOM_D | To calculate endpoints related to time. |



The Follow-up week4 participants variables will be collected from TB-CAPT-HIV EXULTANT-Week-4-v3 CRF, and the following versions of this document. From this CRF the important variables for the analysis are:

| Variable | | Used in |
|---|---|---|
| label | name | |
| Is the visit taking place? (y/n) | W4_VISIT_YN | To calculate the number of people who come to visit at week 8 |
| Is the visit taking place?, date | W4_VISIT_D | To calculate the time in the study, to draw the study K-M graphs in group of people who come to this visit. |
| If the patient has died, date of death | W4_DEATH_D | To use in the K-M graphs as an endpoint for these participants. |
| Has the patient started TB treatment since discharge? | W4_TB_TX_YN | To calculate the proportion of main study objective |
| Has the patient started TB treatment since discharge?, date | W4_TB_TX_START_D | To calculate the proportion of people started on treatment. |
| Has the patient abandoned TB treatment since last visit? | W4_TB_TX_END_YN | To calculate the failure TB treatment |

The Follow-up week8 participants variables will be collected from TB-CAPT-HIV EXULTANT-Week-8-v3 CRF, and the following versions of this document. From this CRF the important variables for the analysis are:

| | | Used in |
|---|---|---|
| Variabl | е | |
| label | name | |
| Is the visit taking place? (y/n) | W8_VISIT_YN | To calculate the number of people who come to visit at week 8 |



| Is the visit taking place? (date) | W8_VISIT_D | To calculate the time in the study, to draw the study K-M graphs in group of people who come to this visit. |
|---|---|---|
| If the patient has died, date of death | W8_DEATH_D | To use in the K-M graphs as an endpoint for these participants. |
| Has the patient started TB treatment since discharge? | W8_TB_TX_YN | To calculate the proportion of main study objective |
| Has the patient started TB treatment since discharge?, date | W8_TB_TX_START_D | To calculate time at risk |
| Has the patient abandoned TB treatment since last visit? | W8_TB_TX_END_YN | To calculate the failure TB treatment |

From Hospitalization Assessment TB-CAPT-HIV EXULTANT-Hospitalization assessment-v3, and the following versions of this document we will use for the analysis the next variables:

| Variable | | Used in |
|---|---|---|
| label | name | |
| Date of enrolment | ENROL_D | To calculate the participant's start time |
| Time of enrolment (24h format) | ENROL_T | |
| Date of discharge | HOSP_END_D | To calculate the participant's hospitalization |
| Time of discharge (24h format) | HOSP_END_T | time |
| Date of lab result:<br>Sputum Ultra | SP_XP_RES_RECEPT_D | To calculate the time to obtain the laboratory results and classify the |
| Time of lab result:<br>Sputum Ultra | SP_XP_RES_RECEPT_T | primary outcome <= 72h or > 72h for Sputum Ultra sample |



| | I | |
|---|---|---|
| Date of lab result: Urine<br>Ultra | URINE_XP_RES_RECEPT_D | To calculate the time to obtain the laboratory results and classify the |
| Time of lab result: Urine<br>Ultra | URINE_XP_RES_RECEPT_T | primary outcome <= 72h or > 72h for Urine Ultra sample |
| Did the patient have cough during hospitalization? | HOSP_COUGH_YN | We will use to describe symptoms. We will use as a factor |
| | | variable in modelling |
| Did the patient have fever (>38°C) during hospitalization? | HOSP_FEVER_YN | We will use to describe symptoms. |
| nospitalization: | | We will use as a factor variable in modelling |
| Did the patient have night sweats during hospitalization? | HOSP_NIGHT_SWEATS_YN | We will use to describe symptoms. |
| nospitalization: | | We will use as a factor variable in modelling |
| Did the patient lose weight during | HOSP_WEIGHT_LOSS_YN | We will use to describe symptoms. |
| hospitalization? | | We will use as a factor variable in modelling |
| Was TB treatment initiated during hospitalization? | HOSP_TB_TX_YN | To calculate the primary objective variable, start treatment within 72h of enrolment |
| TB treatment initiated, Date and Time | HOSP_TB_TX_START_D<br>HOSP_TB_TX_START_T | |
| If Yes, AND the patient has a microbiologically confirmed TB diagnosis (question 2.3), was the treatment initiated within 72hrs of enrolment? | HOSP_TB_TX_72H_YN | To determine the proportion of microbiologically confirmed TB cases starting treatment within 72 hours |



| If wasn't the treatment initiated within 72hrs of enrolment, reason | HOSP_TB_TX_72H_RSN<br>HOSP_TB_TX_72H_RSN_SPEC | To determine the reasons behind starting treatment failure |
|---|---|---|

The laboratory results we will be collected from (15) TB-CAPT-HIV EXULTANT-LabResults-v3- CRF, and the following version of this document. From this source we will select to study the following variables:

| Varia | ble | Used in |
|---|---|---|
| Label | name | |
| Date of sample collection | SAMP_COL_D | To check the range of dates in context of our research objectives |
| CD4 results | CD4_RES | To analyse the primary objective stratified by this variable |
| Viral load results | VL_RES | To analyse the primary objective stratified by this variable |
| Sputum Xpert Ultra | SP_XP_RES | To determine whether a patient is microbiologically confirmed |
| Urine Xpert Ultra | URINE_XP_RES | To determine whether a patient is microbiologically confirmed |
| Stool Xpert Ultra | STOOL_XP_RES | To determine whether a patient is microbiologically confirmed |
| Xpert Ultra in another specimen I | S1_XP_RES | To determine whether a patient is microbiologically confirmed |
| Xpert Ultra in another specimen II | S2_XP_RES | To determine whether a patient is microbiologically confirmed |

The AlereLAM Results will come from the TB-CAPT-HIV EXULTANT-AlereLAM & CRP v3 form, and the update versions of this document. From this CRF will be get:



| Variable | е | Used in |
|---|---|---|
| Label | name | |
| AlereLAM result | ALERE_RES | To determine whether a patient is microbiologically confirmed To do the sensibility analysis of test |
| If results available, date | ALERE_RES_D | To calculate the lab results time |
| If results available, time | ALERE_RES_T | |
| If results not available, reason | ALERE_RES_YN_RSN | To calculate the proportion and reasons of no AlereLAM result |

The Study Completion participants variables we will collected from TB-CAPT-HIV EXULTANT-StudyCompletion-v3 form, and the following versions of this document. From this CRF the important variables for the analysis are:

| Varia | able | Used in |
|---|---|---|
| Label | name | |
| Did participant complete the study procedures at study visit week 8? | VISIT_WK8_D | To calculate<br>the proportion<br>of endpoints at<br>week 8 |
| Did participant complete the study procedures at study visit week 8? date | VISIT_WK8_D | To calculate<br>the time in the<br>study, to draw<br>the study K-M<br>graphs |
| If not, and the participant withdrew, was withdrawn, dropped out or died during the study, indicate the primary reason | END_RSN | To calculate the proportion deaths, lost to follow-up, withdraws and complete study |



| Date participant completed, | END_D | To calculate |
|----------------------------------|-------|-----------------|
| withdrew, was withdrawn/excluded | | the time in the |
| or dropped out from study, date | | study, to draw |
| | | the study K-M |
| | | graphs |

# 5 Sample Size

We expect the absolute difference in proportions of bacteriological confirmation between the two arms to be 7% (from 19% to 26% from the control to the intervention arm). Sample size was chosen to be sufficient to detect a 36.8% relative increase in the primary outcome in the intervention arm (as compared to the control arm).

Under this premise and the following assumptions:

- Alpha (two sided): 0.05
- Beta (power 80%): 0.2
- Estimated proportions of participants with microbiologically confirmed TB in the control arm 19% and int the intervention arm 26%
- Lost to follow up:5% of recruited participants.

The study will recruit 586 PLHIV participants per trial arm, then we will include in the analysis 1172 participants in total. This number of participants will come from 4 sites (293 participants per arm at each site).

For this calculation we have used the following formulas based on Normal asymptotic approximation for proportions:

Sample Size formula

$$n_{1} = \frac{\left(Z_{1-\mathbf{p},le}\sqrt{(1+\varphi)\overline{p}\left(1-\overline{p}\right)} + Z_{1-\mathbf{p}}\sqrt{\varphi p_{1}\left(1-p_{1}\right) + p_{2}\left(1-p_{2}\right)}\right)^{2}}{\varphi \mid p_{2} - p_{1}\mid^{2}}$$

Power formula



$$\begin{split} \varphi &= \frac{1 - w_1}{w_1} \\ \overline{p} &= \frac{p_1 + \varphi p_2}{1 + \varphi} \\ 1 - \beta &= \Phi \left( \frac{|p_2 - p_1| \sqrt{\varphi n_1} - Z_{1-\varphi n_2} \sqrt{(1 + \varphi)\overline{p}(1 - \overline{p})}}{\sqrt{\varphi p_1(1 - p_1) + p_2(1 - p_2)}} \right) \end{split}$$

#### 6 General Considerations

### 6.1 Timing of Analyses

The analysis will be done after database lock and the data cleaning process is finalized.

We will analyse the data using primarily an intention to treat (ITT) analysis approach. This dataset will be composed for all randomized participants by their assigned intervention independent of participation time of this participants in the study. Also, we will analyse the results using the Per Protocol Population approach.

## 6.1.1 Per Protocol Population

For the primary and some secondary endpoints, we will be using the set of data defined as "per-protocol" (PP). This dataset we will only include participants with all required samples collected and results available within 72 hours from enrolment.

This can shed light on a potential effect of poor adherence to study protocol procedures on the primary and secondary endpoints.

### 6.2 Missing Data

Given the characteristics and design of the trial (including data monitoring activities) we expect a low proportion of missing variables.

We will analyse the mechanisms that cause missing data. We plan to identify the three typical patterns for missing data: missing completely at random (MCAR); missing at random (MAR); and missing not at random (MNAR).

To assess the potential influence of missing values in intervention related variables or visit related variables (due to withdraws or death), we will compare the results of the ITT and per protocol analyses. To assess the potential influence of missing values in endpoint related



variables, we will perform a complete case analysis when the proportion of missing data is below, approximately, 5% and it is implausible that certain patient groups specifically are lost to follow-up in one of the compared arms. In this case we will analyse previously if the missing data are random or follow some pattern.

For missing data over 5%, we will do a worst/best scenario sensitivity analysis for the main endpoint related variables (related TB treatment initiation, time from enrolment and microbiological results). This consists of assigning the best plausible outcome to the above endpoint-related missing values in both arms (i-e TB treatment started, TB treatment started before 72 hours from enrolment, or TB microbiological confirmation) and the other assigning the worst possible outcome to all missing values in both groups (TB treatment not initiated, TB treatment started after 72 hours from enrolment, non-TB microbiological confirmation).

We will also compare the results of one assigning the best possible outcome to missing values in the intervention arm and the worst possible to those of the intervention arm, and vice-versa.

If this sensitivity analyses raise inconsistent results on the intervention effect, their repercussions will be discussed between the statisticians involved in trial analysis.

# 6.3 Multiple Testing

We consider unnecessary to apply a general adjustment of significance level by multiple comparisons test. We will use the all the statistical power for inference only in the primary study objective. To evaluate the other study endpoints, we use the p-value threshold at 0.05 to find the differences in our study without the objective to extrapolate the results to the global community. However, we will establish a p-value of 0.01 as a threshold for statistical significance in the comparisons related to a) selected secondary efficacy analyses (section 8.2, analyses 8.2.5, 8.2.6, 8.2.7) and subgroup analysis (see section 9.0)

We will adjust the results by site, demographic variables, and other baseline variables if we will detect differences or if these variables have a confounder characteristics profile. To decide this, we will do a preliminary analysis of these variables between sites.

# 7 Summary of Study Data

### 7.1 Subject Disposition

We will use the **Study Completion**, **Withdrawal and Drop-out Form** (**TB-CAPT-HIV EXULTANT-StudyCompletion-v3.1**) to show how many participants reached the study stages. Data from this form, **from question 1 to 4**, will allow us to know the number of dropouts and their reasons and how many participants will arrive to week 8 or not.



# 7.2 Derived variables

We will create some derived variables according to solve the study hypothesis, some of them we will describe in the following SAP versions.

The variables that we will create are:

| New Variable | Туре | Values |
|---|---|---|
| Type of Employment | Categorical | 0: Unemployed for any reason |
| | | 1: Health care worker |
| | | 2: Prison warder or work at a correctional facility |
| | | 3: Miner |
| Time from last HIV+ result | Continuous | 0 to randomization date |
| Time of follow-up | Continuous | From randomization date to end study completion date |
| Time to TB treatment initiation | Continuous | From randomization date to start TB treatment date |
| (in hours) | | to start 15 treatment date |
| ITT cohort | Categorical | 0: Not included in ITT |
| | | 1: Included in ITT |
| ATP cohort | Categorical | 0: Not included in ATP |
| | | 1: Included in ATP |
| Participants diagnosed with | Categorical | 0: No |
| microbiologically confirmed TB | | 1: Yes |
| Participants diagnosed with | Categorical | 0: No |
| microbiologically confirmed TB and started on TB | | 1: Yes |
| treatment within 72 hours of enrolment | | |
| CD4 (binary) | Categorical | 0: CD4 count <100 |



| 1: CD4 count >=100 |
|--------------------|

## 8 Efficacy Analyses

# 8.1 Primary Efficacy Analysis

The primary efficacy is defined as the difference in the proportion of microbiologically confirmed TB and therapy initiated within 72 hours from enrolment in the intervention and control arm. (the comparison by estimating the difference of proportions and see whether is significantly differs from zero)

We will compare the difference of proportions, defined above, between both study arms and see if the results are significantly different from zero. We will test this differences using the test statistics z has an asymptotic standard normal distribution, and the p-value will be computed as:

p = 2 {1-  $\Phi$  (|z|)} where  $\Phi$ (·) is the cdf of a standard normal distribution and |z| is an absolute value of z. We will calculate logit-transformed 95% confidence intervals

We will compare this proportion as a risk difference and we will stratify by study countries, baseline CD4 counts (under the hypothesis the highest difference in % of bac confirmed participants between control and intervention arm will occur in those immunosuppressed ones, or in countries with highest % of immunosuppressed admitted participants).

We will evaluate the primary efficacy analysis by ITT and Per protocol populations. We will show the both results in the final analysis document with the correspondent tables and graphs.

# 8.2 Secondary Efficacy Analyses

All secondary efficacy analyses will be calculated on ITT and Per protocol populations. The Secondary Efficacy Analyses are:

8.2.1 We will compare the proportion of deaths during eight weeks after enrolment between all participants enrolled in two study groups. We will test this differences using the test statistics z has an asymptotic standard normal distribution These groups are microbiologically confirmed TB and therapy initiated within 72 hours from admission (numerator/success) and non-lab-confirmed TB or therapy not initiated within 72 hours (denominator/failure). We will compare, using Chi-square test or Fisher Test, these proportion values between intervention and control group.



- 8.2.2 We will estimate the Kaplan Meier curves to assess time to TB treatment initiation among those with microbiologically confirmed TB and among all TB (also including clinically diagnosed). We will compare both arms using the log rank test. We will use the KM procedure to calculate the survival rate from the survival function. If deemed necessary, to study the effects of some covariates and start of treatment over time we will use the Cox regression.
- 8.2.3 We will compare the proportion of cases re-admitted to hospital, to test this proportion we calculate the number of admissions after initial discharge and within 8 weeks from enrolment from all participants enrolled. We will compare, using Chi-square test or Fisher Test, these proportion values between intervention and control group.
- 8.2.4 We will compare the proportion of participants who are diagnosed with TB (irrespective of bacteriological confirmation and are started on TB treatment within 72 hours of enrolment). We will compare, using Chi-square test or Fisher Test, these proportion values between intervention and control group.
- 8.2.5 We will calculate the proportion of participants who are diagnosed with microbiologically confirmed TB and are started on TB treatment at 7d, 14d, 4 and 8 weeks of enrolment. We will compare, using Chi-square test or Fisher Test, these proportion values between intervention and control group.
- 8.2.6 We will calculate the proportion of participants who are able to provide the different samples (sputum and urine) at 24, 48 and 72 hours (or later) from enrolment. We will describe the participants profile for every previous point and participants who are unable to provide these samples. We will compare, using Chi-square test or Fisher Test, these proportion values between intervention and control group.
- 8.2.7 We will analyse the time to laboratory confirmed TB diagnosis and any TB diagnosis since enrolment. For this we will calculate the Kaplan Meier estimator and curves. Additionally, we will do proportional hazards models and calculate the hazard ratios at days 7, 14, 28 and 56 and compare the time related estimates between intervention and control group. The models will use the following covariates from Baseline CRF: Site, Sex, CD4 counts.
- 8.2.8 We will compare the proportion of deaths during first four weeks after enrolment between all participants enrolled in two study groups. We will compare these proportions using Chi-square test or Fisher Test, according to the application condition. These groups are microbiologically confirmed TB and therapy initiated within 72 hours from admission (numerator/success) and non lab-confirmed TB or therapy not initiated within 72 hours (denominator/failure).



8.2.9 We will calculate the proportion of participants started on treatment without Rif resistance information (only AlereLAM positive). We will compare, using Chisquare test or Fisher Test, these proportion values between intervention and control group.

# 9. Subgroup analysis

The analysis of all endpoints will be done for all patients of both countries as sample size did not take into consideration country-specific analyses of the specified primary endpoint. Thus, we will merge the data from the four sites we will analyse the resulting database as unique source of data.

However, a subgroup analysis of the primary endpoint and main secondary endpoint (mortality at month 2) will be done by study site (Mozambique and Tanzania, CD4 counts and viral load).

A separate analysis of the primary and secondary endpoints will also be performed by sex of participants, in order to asses if differences arise in any of the outcomes.

# 10. Other Analyses

We will do a comparison of baseline characteristics between participants who can complete the study and participants who we will lose during their follow-up period. We will do this analysis to test if the participant loss is by chance. We will use Chi2 statistical test. The variables that we will tested are: Country (COUNTRY), Sex (SEX), Ethnic group (ETHNIC), Level of education (EDUCATION), Employment Status (EMPLOYMENT), Early HIV positive result (EARLY\_HIV), Current taking antiretroviral (ART\_YN), Previous TB episodes (TB\_TX\_YN), Received BCG vaccination (BCG\_YN), Participant live alone? (ALONE), Patient taking cotrimoxazole (CTX\_YN), Karnofsky Performance Status Scale (KARNOFSKY), Patient's WHO clinical Stage (WHO\_STAGES) and TB treatment start (TB\_TX\_START\_YN).

# 11 Reporting Conventions

We will use two decimals in numeric results. We will round to up the value of second decimal when the third decimal value will be equal or higher than 5, in other cases we will do nothing.

All confidence intervals (CI) will be calculated at 95% of confidence. These will be calculated using the logit-transformed confidence interval method. We will use the Haybittle-Peto approach for the evaluation of the p-value, under this approach we will consider statistically significant when the p-value's test is lower than 0.05 in the final analysis

Where necessary, variables will be categorized using the cut-off described in previous works and research publish documents. For example, CD4 counts will be categorized in 3: less than 100 CD4 counts per ml (as in STAMP trial), 100-200 CD4 counts per ml, and above 200.



However, depending on the frequencies observed, these categories could be refined. When we don't have a reference cut-off value for a continuous variable, we will calculate these values using the terciles, quartiles or quintiles of the variable and cut it using this calculated cut-off values. (For example, if we want to divide the participants age in three categories, we will calculate the terciles values and later we calculate a new categorical variable using these points. Then we will have a new age group with three categories: from minimum value to first tercile, from first to second tercile and finally from second tercile to maximum value).

#### 12 Technical Details

The statistical analysis we will performed with the Stata software. We will use the Stata 17 version or the most up to date available version when analysis takes place. Scripts used in the analysis can be published as supplementary material of the main publication or uploaded into a public repository.

## 13 Listing of Tables, Listings and Figures

We will show the results using Tables and Figures. The following is a description of these tables. Some of these tables will summarize the results for ITT and per protocol analysis and always we will make it by study arm. According to the figures we will draw the Kaplan-Meier curves to show the proportion of participants initiating TB treatment over time, stratified by lab confirmation, CD4 count category, viral load and country. Venn diagrams showing the distribution of participants starting TB treatment by positivity to each test will be displayed.

Table 1. Baseline Characteristics of participants by study arm for ITT and per protocol analysis

| | | ITT Ar | nalysis | Per Protocol Analysis | |
|---|---|---|---|---|---|
| | | Standard-of- | Intervention | Standard-of- | Intervention |
| | | care group | group | care group | group |
| | | (n=XXXX) | (n=XXXX) | (n=XXXX) | (n=XXXX) |
| Age (years) | | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Gender | | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Country Site | | | | | |
| Moz | ambique | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |



| Tanzania | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
|---|---|---|---|---|
| Employment Status | | | | |
| Employed | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Unemployed | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Unable to work | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Student | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| House man/wife | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Retired | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Other | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Previous TB episodes | | | | |
| Yes | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| No | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| BCG vaccination | | | | |
| Yes | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| No | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Unknown | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Cotrimoxazol treatment | | | | |
| Yes | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| No | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Unknown | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Antiretroviral treatment | | | | |
| Yes | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| No | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Unknown | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| CD4 count <200cells/mm <sup>3</sup> | | | | |
| Yes | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |



| No | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
|--------------------|-----------|-----------|-----------|-----------|
| Who clinical stage | | | | |
| Stage I | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Stage II | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Stage III | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Stage IV | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |

Table 2. Microbiological results by study arm for both the ITT and per protocol analyses

| | I | TT Analysis | | Per | Protocol Analy | /sis |
|---|---|---|---|---|---|---|
| | Standard-<br>of-care<br>group<br>(n=XXXX) | Intervention<br>group<br>(n=XXXX) | p-value | Standard-<br>of-care<br>group<br>(n=XXXX) | Intervention<br>group<br>(n=XXXX) | p-value |
| Samples available | XXX<br>(XX.X) | XX.X<br>(XX.X) | X.XXX | XX.X<br>(XX.X) | XX.X<br>(XX.X) | X.XXX |
| Sputum Ultra available | XXX<br>(XX%) | XXX (XX%) | X.XXX | XXX<br>(XX%) | XXX (XX%) | X.XXX |
| Sputum Ultra results | | | | | | |
| Negative Indeterminate Positive | XXX<br>(XX%)<br>XXX<br>(XX%)<br>XXX<br>(XX%) | XXX (XX%) XXX (XX%) XXX (XX%) | X.XXX | XXX<br>(XX%)<br>XXX<br>(XX%)<br>XXX<br>(XX%) | XXX (XX%) XXX (XX%) XXX (XX%) | X.XXX |
| Urine Ultra available | | XXX (XX%) | | | XXX (XX%) | |
| Urine Ultra results | | | | | | |
| Negative | | XXX (XX%) | | | XXX (XX%) | |
| Indeterminate | | XXX (XX%) | | | XXX (XX%) | |



| Positive | | XXX (XX%) | | | XXX (XX%) | |
|---|---|---|---|---|---|---|
| Stool Ultra available | | XXX (XX%) | | | XXX (XX%) | |
| Stool Ultra results | | | | | | |
| Negative | | XXX (XX%) | | | XXX (XX%) | |
| Indeterminate | | XXX (XX%) | | | XXX (XX%) | |
| Positive | | XXX (XX%) | | | XXX (XX%) | |
| AlereLAM available | XXX<br>(XX%) | | | XXX<br>(XX%) | | |
| AlereLAM results | | | | | | |
| Negative<br>Indeterminate<br>Positive | XXX<br>(XX%)<br>XXX<br>(XX%)<br>XXX<br>(XX%) | | | XXX<br>(XX%)<br>XXX<br>(XX%)<br>XXX<br>(XX%) | XXX (XX%) XXX (XX%) XXX (XX%) | |
| Microbiologically confirmed | XXX<br>(XX.X) | XX.X<br>(XX.X) | X.XXX | XX.X<br>(XX.X) | XX.X<br>(XX.X) | X.XXX |

Table 3. TB treatment initiation within 72 hours

| | ITT Analysis | | | Per Protocol Analysis | | |
|---|---|---|---|---|---|---|
| | Standard-of-<br>care group | Intervention<br>group | p-value | Standard-of-<br>care group | Intervention<br>group | p-value |
| | (n=XXXX) | (n=XXXX) | | (n=XXXX) | (n=XXXX) | |
| Start treatment within 72 hours | XXX (XX.X%) | XXX (XX.X%) | X.XXX | XXX (XX.X%) | XXX (XX.X%) | X.XXX |
| Hours to start treatment (treatments <= 72h) | XXX (XX%) | XXX (XX%) | X.XXX | XXX (XX%) | XXX (XX%) | X.XXX |



# **Statistical Analysis Plan**

| Days to start<br>treatment<br>(treatments ><br>72h) | XXX (XX%) | XXX (XX%) | X.XXX | XXX (XX%) | XXX (XX%) | X.XXX |
|---|---|---|---|---|---|---|
| Start treatment within 72 hours | | | | | | |
| Confirmed TB | XXX (XX%) | XXX (XX%) | X.XXX | XXX (XX%) | XXX (XX%) | X.XXX |
| Unconfirmed<br>TB | XXX (XX%) | XXX (XX%) | X.XXX | XXX (XX%) | XXX (XX%) | X.XXX |

# Table 4 TB outcomes at 8 weeks by arm (ITT analysis)

| | Standard-of- | Intervention | | |
|---|---|---|---|---|
| | care group | group | Risk Difference | p-value |
| | (n=XXXX, %) | (n=XXXX, %) | % (95% CI) | |
| Start treatment within 72 hours | XXX (XX.X) | XX.X (XX.X) | X.X (X.X, X.X) | X.XXX |
| Microbiologically confirmed TB | XXX (XX%) | XXX (XX%) | X.X (X.X, X.X) | X.XXX |
| Clinically diagnosed TB | XXX (XX%) | XXX (XX%) | X.X (X.X, X.X) | X.XXX |
| Deaths at week 8 | XXX (XX%) | XXX (XX%) | X.X (X.X, X.X) | X.XXX |



Figure 1. Trial flowchart

